CLINICAL TRIAL: NCT00481442
Title: Effects of Phenylephrine on Systemic and Regional Hemodynamics in Patients With Septic Shock: a Crossover Pilot Study
Brief Title: Phenylephrine Versus Norepinephrine in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1125
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-03

CONDITIONS: Septic Shock
Keywords: Septic shock; Sepsis; Norepinephrine; Phenylephrine
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Phenylephrine

SUMMARY:
Clinical studies evaluating the clinical use of phenylephrine in septic shock are lacking. The present study was designed to compare the effects of norepinephrine and phenylephrine on systemic and regional hemodynamics in patients with catecholamine-dependent septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Clical diagnosis of Septic Shock
* norepinephrine to maintain mean arterial pressure between 65 and 75 mmHg despite adequate volume resuscitation (pulmonary artery occlusion pressure = 12-18 mmHg and central venous pressure = 8-12 mmHg).

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Present or suspected acute coronary artery disease
* Present or suspected acute mesenteric ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Systemic and regional hemodynamics | 24 hours

SECONDARY OUTCOMES:
Organ functions, adverse effects | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Morelli, MD, Principal Investigator — Departement of Anesthesiology and Intensive Care of the University of Rome "La Sapienza"
Locations (1):
- Department of Anesthesiology and Intensive care of the University of Rome "La Sapienza", Rome, Italy